CLINICAL TRIAL: NCT06622499
Title: Rapid Intravenous Infusion of 10 and 22 Degrees Celsius Ringer's Lactate in Healthy Volunteers and Its Effects on Circulation and Hemostasis - a Randomized Crossover Trial
Brief Title: The Colder Fluids - Intravenous Infusion of 10 Degrees Celsius Fluids and Its Effects on Circulation and Hemostasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506018-35-00
Record Dates: First submitted 2024-06-17; First posted 2024-10-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold - Room temperature (Active Comparator): Trial day 1: Participants receive Ringer's lactate cold (10°C, 50°F), Trial day 2: Participants receive Ringer's lactate at room temperature (22°C, 71.6°F)
  Interventions: Drug: Ringer's Lactate
- Room temperature - Cold (Active Comparator): Trial day 1: Participants receive Ringer's lactate at room temperature (22°C, 71.6°F), Trial day 2: Participants receive Ringer's lactate cold (10°C, 50°F)
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Ringer's Lactate — On the first trial day healthy volunteers are randomized to receive 1 liter of Ringer's lactate either cold (10°C, 50°F), or at room temperature (22°C, 71.6°F) with 100 ml/min. After a minimum "washout period" of 24 hours, subjects are switched to receive infusion at the other aforementioned temperatures.

SUMMARY:
The aim of this study is to investigate the effect of respectively 10 and 22 degrees Celsius Ringer's lactate solution on the physiological response in healthy adults. In a single center crossover study the investigators will include and randomize 25 healthy volunteers to receive 1 liter of Ringer's lactate either cold (10°C, 50°F), or at room temperature (22°C, 71,6°F) with 100 ml/min. Fluids will be administered through a peripheral vein. After a minimum "washout period" of 24 hours, subjects are switched to receive infusion at the other aforementioned temperatures.

The main outcomes of this study are:

Primary:

• The increase in Mean Arterial Pressure (MAP) 30 minutes after started infusion

Secondary:

* Time until return of MAP to baseline value after infusion.
* Changes in Visual Analog Scale (VAS) of discomfort during infusion
* Changes in temperature, blood pressure, heart rate, peripheral oxygen saturation cardiac index, cardiac output, total peripheral resistance index and stroke volume
* Changes in the intravascular volume status and the fluid responsiveness
* Changes in biochemical parameters at baseline, 30 and 60 minutes.
* Changes in Rotational thromboelastometry (ROTEM) analysis at baseline, 30 and 60 minutes

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64

Exclusion Criteria:

* Pre-existing medical problems that are contraindicated for cold crystalloid infusions.
* Pregnancy (validated through a certified urine pregnancy test)
* Body mass index >35 kg/m2
* Medication use, including over-the-counter anti-pyretics within 48 hours, with exception of allergy medication and contraceptives.
* Any family history or predisposition of coagulopathies.
* Any intake of inhibitors of 11β-Hydroxysteroid dehydrogenase the past 48 hours (products containing liquorice)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Increase in Mean Arterial Pressure (MAP) 30 minutes after started infusion | Trial day 1 & Trial day 2

SECONDARY OUTCOMES:
Time until return of Mean Arterial Pressure (MAP) to baseline value after infusion | Trial day 1 & Trial day 2
Changes in Visual Analog Scale (VAS) of discomfort during infusion | Trial day 1 & Trial day 2
  Visual analoge scale of discomfort to assess participants discomfort during the trial. A scale labelled from 0=no discomfort to 10=maximum discomfort imaginable.
Changes in physiological parameter temperature measured in degrees Celcius | Trial day 1 & Trial day 2
Changes in physiological parameter blood pressure measured in millimeter of mercury (mmHg) | Trial day 1 & Trial day 2
Changes in physiological parameter peripheral oxygen saturation measured in percent (%) | Trial day 1 & Trial day 2
Changes in physiological parameter cardiac index measured in L/min/m2 | Trial day 1 & Trial day 2
Changes in physiological parameter cardias output measured in L/min | Trial day 1 & Trial day 2
Changes in physiological parameter total peripheral resistance index measured in dyn·s/cm5 | Trial day 1 & Trial day 2
Changes in physiological parameter stroke volume measured in mL | Trial day 1 & Trial day 2
Changes in physiological parameter intravascular volume status and fluid responsiveness measured in vena cava inferior maximum diameter and index via ultrasound | Trial day 1 & Trial day 2
Changes in physiological parameter of INR blood test measured in prothrombin time at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2
Changes in physiological parameter APTT blood test measured in seconds at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2
Changes in physiological parameter Fibrinogen blood test measured in µmol/L at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2
Changes in physiological parameter Platelet count blood test measured in 109/L at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2
Changes in physiological parameter Flowcytometry blood tests (CD63, CD62p, PAC-1) measured in % at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2
Changes in physiological parameter Rotational thromboelastometry (EXTEM, INTEM, FIBTEM analysis of Clotting time and maximum clot formation) measured in seconds and millimeters, respectively, at baseline, after 30 minutes and after 60 minutes | Trial day 1 & Trial day 2

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Brabrand, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No